CLINICAL TRIAL: NCT01229059
Title: Assessment of the Time Course of Lipid Induced Insulin Resistance
Brief Title: Free Fatty Acid Induced Insulin Resistance
Acronym: FFAIR
Status: Completed | Type: Observational
Sponsor: German Diabetes Center (Other)
Collaborators: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: FFAIR
Record Dates: First submitted 2010-03-20; First posted 2010-10-27 (Estimated); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Insulin Resistance
Keywords: FFA; insulin resistance; mitochondria
MeSH Terms: conditions — Insulin Resistance | interventions — Soybean Oil

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — muscle biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- lipid infusion in untrained humans: healthy lean humans before and after lipid infusion
  Interventions: Dietary Supplement: Lipovenös lipid infusion
- lipid infusion in athletes: endurance trained atheletes
  Interventions: Dietary Supplement: Lipovenös lipid infusion

INTERVENTIONS:
Dietary Supplement: Lipovenös lipid infusion — Lipid enriched infusions will be applied for 2-6 hours.
  Other Names: soy oil

SUMMARY:
This study aims to explore time-dependent effects of lipid infusion an intramyocellular lipid metabolites and the induction of impaired insulin signaling.

DETAILED DESCRIPTION:
Increased availability of free fatty acids impairs glucose disposal in young healthy humans. Patients with type 2 diabetes have reduced whole body glucose disposal, increased ectopic lipid deposition in skeletal muscle and the liver and impaired mitochondrial function. Recent studies suggest that lipid metabolites such as diacylglycerol (DAG), ceramides and long-chain acyl-coA represent the active mediators inducing insulin resistance. Possible targets are DAG-sensitive Proteinkinase C (PKC θ, PKC ε) which inhibit the insulin signaling cascade and ceramides which interfere with the insulin signaling cascade at Proteinkinase B/AKT. Prior studies raised controvesial evidence, thus, it is yet unclear, whether DAG or ceramides are the primary agents inducig lipid-induced insulin resistance. Therefore, the current study aims to explore the time course of the appearance of intramyocellular lipid compunds during lipid infusion in parallel assessing markers of impaired insulin action.

ELIGIBILITY:
Inclusion Criteria:

* non-diabetic (OGTT), no family history of diabetes, BMI<30 kg/m2, age: 20-55 years, no medication

For the athletes group additionally:

* VO2max > 60ml/kg/min for males and VO2max > 45ml/kg/min for females Active in endurance-exercise activities, 3 times a week for at least 2 years Stable level of training for at least 3 months

Exclusion Criteria:

* acute illness within the last 2 weeks, autoimmune diseases, renal insufficiency (creatinine> 1.5 mg/dl), cardiovascular diseases, anemia (Hb< 12g/l), donation of blood within the last 4 weeks before the study, thyroid diseases, pregnancy, smoking, night-shift working (disturbed circadian rhythm), defective coagulation or wound healing, cancer, allergy against soja products

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, lean non-diabetic humans
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
intramyocellular lipid metabolites | after 4 hours lipid infusion
  Muscle biopsies are taken before, after 2.5 and 4 hours of lipid infusion
muscle glucose flux | during lipid infusion
  glycogen synthesis rate, glucose-6-phosphate

SECONDARY OUTCOMES:
insulin resistance of glucose uptake and mitochondrial function | after 4 hours lipid infusion
  Mitochondrial function will bes assessed from muscle biopsy samples taken after 4 hours, insulin sensitivity will be assessed from hyperinsulinemic-euglycemic clamps following 4 hours lipid infusion

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Prof., MD, Principal Investigator — German Diabetes Center
Locations (1):
- German Diabetes Center, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Phielix E, Begovatz P, Gancheva S, Bierwagen A, Kornips E, Schaart G, Hesselink MKC, Schrauwen P, Roden M. Athletes feature greater rates of muscle glucose transport and glycogen synthesis during lipid infusion. JCI Insight. 2019 Nov 1;4(21):e127928. doi: 10.1172/jci.insight.127928. PMID 31672941
- [Derived] Fritsch M, Koliaki C, Livingstone R, Phielix E, Bierwagen A, Meisinger M, Jelenik T, Strassburger K, Zimmermann S, Brockmann K, Wolff C, Hwang JH, Szendroedi J, Roden M. Time course of postprandial hepatic phosphorus metabolites in lean, obese, and type 2 diabetes patients. Am J Clin Nutr. 2015 Nov;102(5):1051-8. doi: 10.3945/ajcn.115.107599. Epub 2015 Sep 30. PMID 26423389